CLINICAL TRIAL: NCT03561064
Title: Improving Sleep in Cancer Patients: A Feasibility Trial of Implementing Cognitive Behavioral Therapy for Insomnia During Cancer Treatments
Brief Title: Improving Sleep in Cancer Patients: A Feasibility Trial
Acronym: ISCAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Sivan Rotenberg, Assistant Professor, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D18087
Record Dates: First submitted 2018-05-25; First posted 2018-06-19 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Cancer; Insomnia
Keywords: cancer; insomnia; CBT; CBT-I; cognitive behavioral therapy
MeSH Terms: conditions — Neoplasms; Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Receiving CBT-I (Experimental): This is a single arm study. All participants will receive CBT-I (cognitive behavioral therapy for insomnia).
  Interventions: Behavioral: CBT-I

INTERVENTIONS:
Behavioral: CBT-I — Eligible participants will receive CBT-I by a licensed clinical psychologist.
  Other Names: cognitive behavioral therapy for insomnia

SUMMARY:
The purpose of this study is to determine if CBT-I (cognitive behavioral therapy for insomnia) is a feasible treatment for insomnia in individuals undergoing cancer treatment.

DETAILED DESCRIPTION:
This research study is a single arm feasibility trial in which all eligible participants receive five weekly sessions of CBT-I (cognitive behavioral therapy for insomnia) delivered before or during their cancer treatments. CBT-I is a non-drug behavioral treatment for insomnia and is considered the most effective treatment for insomnia. However, CBT-I is not routinely offered to cancer patients due to unknowns about its feasibility in this population. Data will be obtained at pre- and post-CBT-I and at eight-week follow-up, and will focus on acceptability, implementation, and efficacy in order to assess feasibility. The study will focus on cancer patients who are diagnosed with gastro-intestinal (GI) cancer.

ELIGIBILITY:
Inclusion Criteria:

1. 18+ years of age
2. have insomnia disorder (SOL or WASO greater than 30 minutes for more than 6 nights in two weeks + daytime impairments)
3. are diagnosed with gastro-intestinal cancer;
4. have life expectancy > 6 months;
5. are fully ambulatory indicated by the provider-rated score of greater than 2 on the Eastern Cooperative Oncology Group (ECOG) performance measure;
6. will complete cancer treatments in no less than seven weeks, allowing for two weeks of assessments and five weeks of CBT-I;
7. are English-speaking and able to provide voluntary, written consent.

Exclusion Criteria:

1. unmanaged sleep apnea indicated by the scores on the STOP-BANG Questionnaire suggesting high risk for sleep apnea and not receiving any sleep apnea treatment;
2. other sleep disorders;
3. bipolar disorder;
4. unmanaged serious mental illnesses;
5. suicidal ideation/intent/plan;
6. unstabilized pharmacological treatment for insomnia;
7. night-shift employment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Change of the score on the Insomnia Severity Index (ISI) | baseline and at 19th week
  The ISI assesses the severity of insomnia symptoms and subjective daytime impairments.

SECONDARY OUTCOMES:
Change of diary-assessed sleep onset latency | baseline and at 19th week
  Sleep onset latency is the time it takes to fall asleep
Change of diary-assessed wake after sleep onset | baseline and at 19th week
  wake after sleep onset is the total duration of nighttime awakenings
Change of actigraphy-sleep onset latency | baseline and at 19th week
  Sleep onset latency is the time it takes to fall asleep
Change of actigraphy-assessed wake after sleep onset | baseline and at 19th week
  wake after sleep onset is the total duration of nighttime awakenings

CONTACTS AND LOCATIONS:
Overall Officials: Wai S Chan, PhD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.